CLINICAL TRIAL: NCT05660616
Title: Switch-Maintenance Gemcitabine After First-Line Chemotherapy (Pemetrexed-Platinum) In Patients With Malignant Pleural Mesothelioma In Ain Shams University Hospitals
Brief Title: Switch-Maintenance Gemcitabine After First-Line Chemotherapy In Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMGFM
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-02

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Mesothelioma; Switch-maintenance; Gemcitabine
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Gemcitabine; Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gemcitabine + supportive care (Experimental): Administration of maintenance gemcitabine (1000 mg/m²) on days 1 and day 8, in cycles of 21 days plus supportive care.
  Interventions: Drug: Gemcitabine; Other: supportive care
- supportive care (Other): best supportive care alone.
  Interventions: Other: supportive care

INTERVENTIONS:
Drug: Gemcitabine — The study includes patients with unresectable malignant pleural mesothelioma who received at least 4 cycles of first line platinum (Cisplatin or Carboplatin) and pemetrexed combination chemotherapy
  * Response after first line treatment will be assessed by the modified Response Evaluation Criteria in Solid Tumors (mRECIST) version 1.1 for pleural mesothelioma.
  * Patients will be randomized according to a (1:1) ratio to either Arm 1: Administration of maintenance gemcitabine (1000 mg/m²) on days 1 and day 8, in cycles of 21 days plus supportive care Arm 2 (control arm): best supportive care alone.
  * Cases will be evaluated every cycle clinically and every three cycles radiologically with CTs.
  Other Names: Gemzar
  Arms: Gemcitabine + supportive care
Other: supportive care — supportive care

SUMMARY:
Mesothelioma is an aggressive form of cancer. Treatments are available, but for many people, a cure isn't possible.

This thesis is to assess the efficacy and safety of switch-maintenance Gemcitabine in Mesothelioma patients after first line chemotherapy (Pemetrexed-Platinum)

DETAILED DESCRIPTION:
Malignant pleural mesothelioma is a rare but aggressive cancer of the pleural lining.

Malignant pleural mesothelioma accounted for 30,870 new cancer cases and 26,278 deaths worldwide in 2020.

In Egypt, Malignant pleural mesothelioma accounted for 337 new cases and 307 deaths in 2020.

Long-term exposure to asbestos is a well-established risk factor for Malignant pleural mesothelioma. It accounts for almost 80% of cases.

Malignant pleural mesothelioma is classified into three histologic subtypes: epithelioid, sarcomatoid, and biphasic. Epithelioid histology confers the most favorable prognosis and sarcomatoid the least.

The majority of patients with Malignant pleural mesothelioma present with breathlessness, chest pain or both. Other symptoms include fatigue, anorexia, weight loss, sweats and malaise.

Radiological imaging should be undertaken in all patients as it can provide valuable diagnostic and staging information. Further investigation of suspected Malignant pleural mesothelioma requires sampling of pleural fluid for biochemical and cytological examination. Biopsies are usually required to confirm the diagnosis and identify the histological sub-type.

Patients with Malignant pleural mesothelioma should be managed by an experienced multidisciplinary team. Treatment options include surgery, radiation therapy and chemotherapy.

Front line polychemotherapy is considered the standard of care, whereas single agent chemotherapy has shown limited efficacy with disappointing response rates.

A pivotal trial led to the establishment of Cisplatin and Pemetrexed as standard first line regimen for unresectable Malignant pleural mesothelioma.

A recent phase II trial from Cancer and Leukemia Group B showed that maintenance Pemetrexed after 4 to 6 cycles of doublet chemotherapy induction did not prolong progression free survival over placebo.

Adding Bevacizumab to first line platinum doublet resulted in an overall survival and progression free survival gain in the phase III French trial MAPS .Bevacizumab was continued as maintenance every three weeks following completion of six cycles of chemotherapy.

In a phase III trial NVALT 5 , Thalidomide versus active supportive care for maintenance in patients with malignant mesothelioma after first-line chemotherapy showed no benefit in time to progression.

First line Nivolumab plus Ipilimumab in phase III trial checkmate 743 provided significant and clinically meaningful improvements in overall survival versus standard of care chemotherapy.

Unfortunately, nearly all patients progress during or after first-line therapy, and no standard second line recommended treatments exist after platinum based regimen. Retreatment with pemetrexed, eventually associated with platinum compound, may be offered in patients who achieved durable disease control more than 6 months with first line chemotherapy.

Single agent chemotherapy with Vinorelbine or Gemcitabine is the preferred choice as second line treatment , mainly based on retrospective analyses or small phase II trials.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Histologically or cytologically confirmed unresectable malignant pleural mesothelioma
* ECOG Performance status 0-2
* Completed at least four cycles of first line platinum (cisplatin or carboplatin) and pemetrexed combination chemotherapy before study entry
* No evidence of disease progression following first-line treatment based on radiological criteria.
* Adequate organ function is mandatory, defined as haemoglobin of at least 8.5 mg/dl, platelets of at least 100×10⁹ per L, and neutrophils of at least 1×10⁹/L.

Exclusion Criteria:

* Progression of disease after first line
* Pregnant females
* ECOG Performance 3-4
* Patients with sarcomatoid mesothelioma
* Patients who are candidates for curative surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
progression free survival | 2 years
  It is the time from randomization to disease progression or death from any cause

SECONDARY OUTCOMES:
overall survival | 2 years
  It is the time from randomization to death from any cause
Toxicity of chemotherapy | 2 years
  toxicity of chemotherapy using CTCAE-version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Abanoub Samir, Principal Investigator — Assistant Lecturer
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karam AS, Abdelwahab S, Ezz El Din MMA, Alorabi MO. A randomized comparative study on maintenance gemcitabine versus supportive care in pleural mesothelioma. Future Oncol. 2025 Jul;21(17):2203-2213. doi: 10.1080/14796694.2025.2516412. Epub 2025 Jun 12. PMID 40501447